CLINICAL TRIAL: NCT06764537
Title: Evaluation of in Vitro Antitumor Activity of GD2 CAR-T Cells Generated From Blood of Glioblastoma Patients
Brief Title: Evaluation of in Vitro Antitumor Activity of GD2 CAR-T Cells in Glioblastoma
Acronym: BOOSTCAR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, REPPEL Loïc, Associate Professor, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RIPH2: 2024-A02098-39 2022PI15
Record Dates: First submitted 2024-11-28; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; GD2 CAR-T cells; Myeloid-derived suppressor cells; microenvironment
MeSH Terms: conditions — Glioblastoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood collection (40 mL) of glioblastoma patients (Experimental)
  Interventions: Procedure: Blood collection

INTERVENTIONS:
Procedure: Blood collection — Blood collection (40 mL) in glioblastoma patients

SUMMARY:
Glioblastoma is a brain tumor with a very poor prognosis, affecting around 2,400 new patients every year. Current treatments do not provide good control of the disease. In view of the therapeutic impasse, it is necessary to develop new strategies. CAR-T cells (Chimeric antigen receptor T cells) represent a highly promising therapy for the treatment of incurable cancers, including glioblastoma. This treatment aims to destroy cancer cells by relying on the patient's own immune system. CAR-T cells are generated from the patient's own immune cells, more specifically T lymphocytes, which are genetically modified to express a tumor-specific receptor on their surface. CAR-T cells bind to tumor cells and cause their destruction. However, these cells have shown limited therapeutic power in the treatment of brain tumors. This is mainly due to the microenvironment surrounding the tumor, which is composed of immunosuppressive cells. These cells, and the molecules they secrete, help to reduce the activity of CAR-T cells that would otherwise reach the tumor. Little is currently known about these resistance mechanisms. The aim of this research is therefore to better understand these resistance mechanisms in order to propose a strategy for enhancing the therapeutic action of CAR-T cells in the treatment of glioblastoma.

The main objective of this research is to evaluate the impact of the tumor environment on the antitumor efficacy of anti-GD2 CAR-T therapeutic cells in an in vitro glioblastoma model. Both tumor environment cells and CAR-T therapeutic cells will be generated from glioblastoma patient cells.

The secondary objectives of this research are to

* Evaluate the impact of tumor environment targeting on the in vitro antitumor efficacy of anti-GD2 CAR-T therapeutic cells.
* Evaluate the quality/quantity of generated cells (CAR-T cells and tumor environment cells) in relation to glioblastoma patients.
* Evaluate the efficiency of the cell isolation technique (CAR-T cells and tumor environment cells)

ELIGIBILITY:
Inclusion Criteria:

* Male or female, adult (age ≥ 18 years)
* WHO 0 to 2
* Patient with a diagnosis of histologically proven de novo glioblastoma with non-mutated IDH status according to WHO 2021 classification
* Patient naïve to any treatment for this cancer
* Patient weighing ≥ 50 kg
* Patient able and willing to follow all study procedures in accordance with the protocol;
* Person affiliated to a social security scheme or beneficiary of such a scheme
* Person who has received full information on the organization of the clinical research and has signed an informed consent form

Exclusion Criteria:

* People with hematological malignancies
* People with a history of cancer < 5 years old
* Immunocompromised (with immunodeficiency or current immunosuppressive therapy)
* Chronic inflammatory disease
* Person with current infection
* Anyone taking corticosteroids >10mg/day on the day of blood sampling for research purposes
* Anyone with a contraindication to blood sampling
* Women of childbearing age without effective contraception
* Persons covered by articles L. 1121-5, L. 1121-7 and L1121-8 of the French Public Health Code Pregnant, parturient or breast-feeding women Minor (not emancipated) Adult subject to a legal protection measure (guardianship, curatorship, safeguard of justice) Persons of full age who are unable to give their consent
* Persons deprived of their liberty by a judicial or administrative decision, persons under psychiatric care under articles L. 3212-1 and L. 3213-1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Quantification of the number of residual tumor cells after in vitro co-culture in presence of CAR-T and MDSC cells | 14 days after the blood sample realized at the inclusion visit
  Using in vitro cytotoxicity tests
The percentage of proliferative effector cells | 14 days after the blood sample realized at the inclusion visit
  Using flow cytometry
The quantity of cytokines released | 14 days after the blood sample realized at the inclusion visit
  Using ELISA tests

CONTACTS AND LOCATIONS:
Locations (1):
- Cell Therapy Unit, Nancy Hospital, Vandœuvre-lès-Nancy, France